CLINICAL TRIAL: NCT06012136
Title: A Phase 1 Double-Blind (Sponsor-unblinded), Placebo-Controlled, Randomized, Single Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of a Parenterally Administered Suspension of Investigational Capsid Inhibitors in Healthy Adults
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of a Single Suspension Injection of Investigational Capsid Inhibitors Compared to Placebo in Healthy Adults
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 218306
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: HIV Infections
Keywords: Healthy participants; Human Immunodeficiency Virus (HIV-1); VH4004280; VH4011499; Long-Acting Injection; Single ascending dose
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Part 1 Single Ascending Dose (SAD): Participants Receiving VH4004280 (Experimental): VH4004280 injections are administered subcutaneously (SC), SC+ rHuPH20, or intramuscularly (IM).
  Interventions: Drug: VH4004280
- Part 1: Participants Receiving Placebo (Placebo Comparator): Placebo injection is administered.
  Interventions: Drug: Placebo
- Part 2 SAD: Participants Receiving VH4011499 (Experimental): VH4011499 injections are administered SC, SC+ rHuPH20, or IM.
  Interventions: Drug: VH4011499
- Part 2 Multiple Ascending Dose (MAD): Participants Receiving VH4011499 (Experimental): VH4011499 injections are administered IM.
  Interventions: Drug: VH4011499
- Part 2: Participants Receiving Placebo (Placebo Comparator): Placebo injection is administered.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VH4004280 — VH4004280 will be administered.
  Arms: Part 1 Single Ascending Dose (SAD): Participants Receiving VH4004280
Drug: Placebo — Placebo will be administered.
  Arms: Part 1: Participants Receiving Placebo; Part 2: Participants Receiving Placebo
Drug: VH4011499 — VH4011499 will be administered.
  Arms: Part 2 Multiple Ascending Dose (MAD): Participants Receiving VH4011499; Part 2 SAD: Participants Receiving VH4011499

SUMMARY:
The primary purpose of the study is to investigate safety and tolerability following single and multiple ascending subcutaneous (SC) and intramuscular (IM) doses of capsid inhibitors in healthy participants. The study will also describe the pharmacokinetics following single and multiple ascending SC and IM doses of capsid inhibitors in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy.
* Participants who are negative on a single test for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) (approved molecular polymerase chain reaction (PCR), point of care test), performed on the day of admission (Day -1). A negative result is required prior to the administration of study intervention on Day 1.
* Male or female participants of non-childbearing potential.
* Capable of giving signed informed consent.

Exclusion Criteria:

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, neurological or psychiatric disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention or interfering with the interpretation of data.
* Abnormal blood pressure.
* Lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Breast cancer within the past 10 years.
* Current or chronic history of liver disease or known hepatic or biliary abnormalities.
* History of sensitivity to any of the study interventions, a history of drug allergy or other allergy that contraindicates their participation.
* The participant has an underlying skin disease or disorder that would interfere with assessment of injection sites.
* Participants considered to have insufficient musculature to allow safe capsid inhibitor intramuscular (gluteus medius) administration.
* History of or on-going high-risk behaviours that may put the participant at increased risk for HIV.
* Past or intended use of over-the-counter or prescription medication including herbal medications.
* Current enrollment or recent past participation in another investigational study.
* Exposure to more than 4 investigational products within 12 months prior to dosing.
* Alanine transaminase (ALT) ≥1.5x upper limit of normal (ULN), Total bilirubin ≥1.5x ULN (isolated total bilirubin >1.5xULN), and/or estimated creatinine clearance (eGFR) of <60 millilitre per minute (mL/min)/1.73 square meter (m^2).
* History of or current infection with hepatitis B or hepatitis C.
* Positive SARS-CoV-2 polymerase chain reaction test, having signs and symptoms, or having contact with known coronavirus disease 2019 (COVID-19) positive person/s in the 14 days prior to inpatient admission.
* Use of tobacco or nicotine-containing products, regular alcohol consumption and/or regular use of known drugs of abuse.
* Positive HIV antibody/antigen test.
* Abnormal electrocardiogram (ECG) parameters.
* Evidence of previous myocardial infarction, any conduction abnormality, any significant arrhythmia, non-sustained or sustained ventricular tachycardia, and/or sinus pauses (>3 seconds).
* The participant has a tattoo or other dermatological condition overlying the location of injection or a prior history of silicone implants or fillers (gluteal) which may interfere with interpretation of injection site reactions or administration of study product.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2023-08-24 (Actual); Primary Completion 2026-06-09 (Estimated); Study Completion 2026-06-09 (Estimated)

PRIMARY OUTCOMES:
SAD: Number of Participants with Adverse Events (AEs) as per Severity | Up to Week 52
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Severity of Adverse Event will be assessed using Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS). DAIDS grading scale is used to grade the toxicity associated with injection site reactions (ISR) including injection site pain (or tenderness), erythema (or redness), induration (or swelling), and pruritis. The toxicity level is graded from grade 1(lowest toxicity) to 4 (highest toxicity). Higher grade indicates higher toxicity.
MAD: Number of Participants with Adverse Events (AEs) as per Severity | Up to Week 56
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Severity of Adverse Event will be assessed using Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS). DAIDS grading scale is used to grade the toxicity associated with injection site reactions (ISR) including injection site pain (or tenderness), erythema (or redness), induration (or swelling), and pruritis. The toxicity level is graded from grade 1(lowest toxicity) to 4 (highest toxicity). Higher grade indicates higher toxicity.
SAD: Absolute Values of Liver Chemistry Parameters: Total Bilirubin and Direct Bilirubin (micromoles per liter [umol/L]) | Up to Week 52
MAD: Absolute Values of Liver Chemistry Parameters: Total Bilirubin and Direct Bilirubin (micromoles per liter [umol/L]) | Up to Week 56
SAD: Change from Baseline in Liver Chemistry Parameters: Total Bilirubin and Direct Bilirubin (umol/L) | Baseline (Prior to Day 1) and up to Week 52
MAD: Change from Baseline in Liver Chemistry Parameters: Total Bilirubin and Direct Bilirubin (umol/L) | Baseline (Prior to Day 1) and up to Week 56
SAD: Number of Participants with Maximum Toxicity Grade Change from Baseline in Liver Chemistry Parameters: Total Bilirubin, Direct Bilirubin, Alkaline Phosphatase, Aspartate Aminotransferase (AST), and Alanine Aminotransferase (ALT) | Up to Week 52
MAD: Number of Participants with Maximum Toxicity Grade Change from Baseline in Liver Chemistry Parameters: Total Bilirubin, Direct Bilirubin, Alkaline Phosphatase, Aspartate Aminotransferase (AST), and Alanine Aminotransferase (ALT) | Up to Week 56
SAD: Absolute Values of Liver Chemistry Parameters: Alkaline Phosphatase, Aspartate Aminotransferase (AST), and Alanine Aminotransferase (ALT) (International Units per liter) | Up to Week 52
MAD: Absolute Values of Liver Chemistry Parameters: Alkaline Phosphatase, Aspartate Aminotransferase (AST), and Alanine Aminotransferase (ALT) (International Units per liter) | Up to Week 56
SAD: Change from Baseline in Liver Chemistry Parameters: Alkaline Phosphatase, AST, and ALT (International Units per liter) | Baseline (Prior to Day 1) and up to Week 52
MAD: Change from Baseline in Liver Chemistry Parameters: Alkaline Phosphatase, AST, and ALT (International Units per liter) | Baseline (Prior to Day 1) and up to Week 56
SAD: Number of Participants with Injection Site Reactions (ISR) AE by Grade Using the DAIDS Grading Scale | Up to Week 52
  DAIDS grading scale is used to grade the toxicity associated with injection site reactions (ISR) including injection site pain (or tenderness), erythema (or redness), induration (or swelling), and pruritis. The toxicity level is graded from grade 1(lowest toxicity) to 4 (highest toxicity). Higher grade indicates higher toxicity.
MAD: Number of Participants with Injection Site Reactions (ISR) AE by Grade Using the DAIDS Grading Scale | Up to Week 56
  DAIDS grading scale is used to grade the toxicity associated with injection site reactions (ISR) including injection site pain (or tenderness), erythema (or redness), induration (or swelling), and pruritis. The toxicity level is graded from grade 1(lowest toxicity) to 4 (highest toxicity). Higher grade indicates higher toxicity.
SAD: Duration of ISR (Days) AE | Up to Week 52
  Duration of ISR will be assessed as the time up to which a reaction related to injection site event is persistent.
MAD: Duration of ISR (Days) AE | Up to Week 56
  Duration of ISR will be assessed as the time up to which a reaction related to injection site event is persistent.
Area Under the Plasma-concentration Time curve from Time Zero to Infinity (AUC0-inf) of VH4004280 | Up to Week 52
Area Under the Plasma-concentration Time curve from Time Zero to Infinity (AUC0-inf) of VH4011499 | Up to Week 56
Maximum Observed Plasma Concentration (Cmax) of VH4004280 | Up to Week 52
Maximum Observed Plasma Concentration (Cmax) of VH4011499 | Up to Week 56
Time of Maximum Observed Plasma Concentration (tmax) of VH4004280 | Up to Week 52
Time of Maximum Observed Plasma Concentration (tmax) of VH4011499 | Up to Week 56
Apparent Terminal Half-life (t1/2) of VH4004280 | Up to Week 52
Apparent Terminal Half-life (t1/2) of VH4011499 | Up to Week 56

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf